CLINICAL TRIAL: NCT02207790
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2609 in Healthy Adult Male Japanese and White Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2609 in Healthy Adult Male Japanese and White Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2609-A001-006
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: Clinical Trial, Phase I; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- E2609 low-dose and placebo in healthy Japanese subjects (Experimental): Cohort 1 will consist of Japanese subjects randomized to a low-dose of E2609 as an orally administered tablet along with subjects receiving matching placebo tablets (matched in number and appearance).
  Interventions: Drug: E2609; Drug: Placebo
- E2609 mid-dose and placebo in healthy Japanese subjects (Experimental): Cohort 2 will consist of Japanese subjects randomized to a mid-dose of E2609 as an orally administered tablet along with subjects receiving matching placebo tablets (matched in number and appearance).
  Interventions: Drug: E2609; Drug: Placebo
- E2609 high-dose and placebo in healthy Japanese subjects (Experimental): Cohort 3 will consist of Japanese subjects randomized to a high-dose of E2609 as an orally administered tablet along with subjects receiving matching placebo tablets (matched in number and appearance).
  Interventions: Drug: E2609; Drug: Placebo
- E2609 mid-dose and placebo in healthy White subjects (Experimental): Cohort 4 will consist of White subjects randomized to a mid-dose of E2609 as an orally administered tablet along with subjects receiving matching placebo tablets (matched in number and appearance).
  Interventions: Drug: E2609; Drug: Placebo

INTERVENTIONS:
Drug: E2609
Drug: Placebo — E2609 low-dose and placebo in healthy Japanese subjects, E2609 mid-dose and placebo in healthy Japanese subjects, E2609 high-dose and placebo in healthy Japanese subjects, E2609 mid-dose and placebo in healthy White subjects

SUMMARY:
This study is primarily designed to bridge the pharmacokinetics (PK) and safety data for E2609 between Japanese subjects and non-Japanese (ie, white) subjects. To bridge these PK characteristics, the proposed study includes a cohort of white subjects treated for comparison with the cohort of Japanese subjects treated at the same dose. This comparison serves as a key PK bridge in assessing ethnic factors that may contribute to differences in plasma concentrations. Pharmacokinetic assessments in the proposed study will include confirmation of dose proportionality in Japanese subjects. This study will also evaluate safety and tolerability in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

The subject must meet all of the following criteria in order to be included in the study.

Japanese Subjects Only:

1. Birth in Japan to Japanese parents and grandparents of Japanese descent
2. Have been living outside Japan for less than 5 years
3. Lifestyle, including diet, has not changed significantly since leaving Japan

   White Subjects Only:
4. A person having origins in any of the original peoples of Europe, the Middle East, or North Africa based on documented subject self-report

   All Subjects:
5. Healthy male, 30 to 60 years inclusive, at the time of informed consent
6. BMI of 18 to 32 kg/m2 inclusive at Screening
7. Subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must not be of childbearing potential or must be practicing highly effective contraception (i.e. condom plus spermicide, condom plus diaphragm with spermicide, intrauterine device starting for at least one menstrual cycle before starting study drug[s]) and throughout the study period and for 30 days after study drug discontinuation. No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

1. Any history of seizures or epilepsy
2. Any medical condition which, in the opinion of the investigator has high risk of seizures
3. Any history of cerebrovascular disease
4. A history of prolonged QTc interval
5. Any other clinically significant ECG abnormalities
6. History of risk factors for torsade de pointes or the use of medications that prolonged the QT/QTc interval
7. Heart rate less than 50 or greater than 100 beats/min
8. History of ischemic heart disease
9. Persistent systolic blood pressure (BP) greater than 140 mmHg or less than 90 mmHg and diastolic BP greater than 90 mmHg or less than 60 mmHg
10. Left bundle branch block
11. Evidence of clinically significant disease
12. Any laboratory abnormalities considered clinically significant
13. Clinically significant illness which requires medical treatment
14. Any history of abdominal surgery that may affect study drugs
15. Hypersensitivity to the study drug
16. Known to be HIV positive
17. Active viral hepatitis
18. History of drug or alcohol dependency or abuse within approximately the last 2 years
19. Scheduled for surgery during the study
20. Engagement in strenuous exercise within 2 weeks before dosing (eg, marathon runners, weight lifters)
21. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days before informed consent

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of E2609: Cmax | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: tmax | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: AUC(0-24h)+D90 | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: AUC(0-72h) | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: AUC(0-t) | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: AUC(0-inf) | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: AUC Metabolite Ratio | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: t1/2 | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: CL/F | Up to Day 10 (216 hours postdose)
Pharmacokinetics of E2609: V/F | Up to Day 10 (216 hours postdose)
To evaluate the safety and tolerability of E2609 | Baseline and up to 30 days from last dosing of subject
  Safety will be assessed by monitoring and recording all adverse events (AEs), serious adverse events (SAEs), regular monitoring of hematology, blood chemistry, urine values, regular measurement of vital signs, ECGs and performance of physical examinations

SECONDARY OUTCOMES:
Pharmacodynamic effect of E2609: percent change from baseline of plasma (AB[1-x]): Amax | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, and Day 10
Pharmacodynamic effect of E2609: percent change from baseline of plasma (AB[1-x]): T(Amax) | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, and Day 10
Pharmacodynamic effect of E2609: percent change from baseline of plasma (AB[1-x]): AUAC(-24h-0h) | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, and Day 10
Pharmacodynamic effect of E2609: percent change from baseline of plasma (AB[1-x]): AUAC(0-144h) | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, and Day 10
Pharmacodynamic effect of E2609: percent change from baseline of plasma (AB[1-x]): Change in AUAC | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, and Day 10
Change from baseline in QTcF obtained from ECGs extracted from Holter recordings | Baseline, Day 1, and Day 2
  Holter ECG measurements will start on Day -1, at a time equivalent to 24 hours predose, and will continue for 24 hours postdose of Day 1, with interruptions allowed to adjust equipment. ECGs will be extracted from Holter monitors.

CONTACTS AND LOCATIONS:
Locations (1):
- Glendale, California, United States